CLINICAL TRIAL: NCT04698733
Title: Efficacy of a Pulsed Microcurrent in the Non-Invasive Treatment of Knee Pain From Osteoarthritis
Brief Title: Veteran Affairs Osteoarthritis Knee Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avazzia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-191011-01-VA-OA-Knee
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
Keywords: electric stimulation; microcurrent; knee pain; knee injury
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: BEST™ Pro-Sport Ultra® microcurrent device (Experimental): Participants will receive 2 treatments a week on nonconsecutive days for 6 weeks in the clinic with an active electrical stimulation device.
  Interventions: Device: BEST™ HVPC microcurrent electrical stimulation Pro-Sport Ultra® device

INTERVENTIONS:
Device: BEST™ HVPC microcurrent electrical stimulation Pro-Sport Ultra® device — Participants will receive two (2) 20-minute treatments a week on nonconsecutive days for 6 weeks in the clinic. At the end of 6 weeks, participants will have a 6-week pause in treatment.
  Active Avazzia PRO-Sport Ultra® medical device, BEST™ HVPC microcurrent electrical stimulation, FDA cleared for pain relief

SUMMARY:
A clinical study at the Dallas Veterans Affairs, is being proposed to test the efficacy of a novel electrical stimulation platform named the Pro-Sport Ultra® device by AVAZZIA to reduce pain and increase activity level in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The primary objective of this study is to document the possible short- and long-term decrease in pain as scored by participants on a Numeric Rating Scale (NRS) after use of Avazzia PRO-Sport Ultra® device with pulsed microcurrent in patients with osteoarthritis of the knee.

Patients with a clinical diagnosis of Osteoarthritis (OA) of the knee for a minimum of 6 months will be recruited for this study. Their OA has not responded/is not responding to treatment and continuing symptoms interfere with normal function. Additionally, patients will have a pain score of 3 or greater on the NRS even with pain medication.

Secondary objectives include changes in:

* Mobility via a Timed Up & Go assessment (TUG). Participants are timed getting up from sitting in a standard armchair, walking approximately 3 meters, turning, walking back to the chair, and sitting down.
* Patient-relevant outcomes via the Knee Injury and Osteoarthritis Outcome Score (KOOS). The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
* Brief Pain Inventory - Short Form
* Use of pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Have a prior diagnosis (Dx) of OA of the knee and have had a trial of conservative treatment for a minimum of 6 months without successful results due to continuing symptoms that interfere with normal function
* Age >18 - <70 years old
* Males/Females of all ethnicities
* NRS pain score of 3 or greater while on medication
* Ability to understand the informed consent document before signing it
* For female participants, is at least 4 years post-menopausal, has a history of hysterectomy, has had bilateral tubal ligation, or consents to use two forms of birth control.

Exclusion Criteria:

* Poor diabetic control (A1c>11 within the last 3 months)
* Diagnosis of acute sciatica and/or acute vasculitis
* Diabetic peripheral neuropathy
* Lower extremity surgery within the last 6 months
* Knee replacement
* Uncontrolled mood disorders, such as depression, anxiety
* Drug or substance abuse within past 90 days
* Injury that results in a change in pain level due to causes other than osteoarthritis (i.e., a recent fall or accident)
* Epilepsy
* Open wounds around knee joint
* Active litigation, workers compensation
* An electrically implanted device such as a pacemaker, neural stimulator, etc.
* Currently pregnant, nursing, or may become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Pain Level Assessment | 12 weeks
  Change in pain associated with osteoarthritis of the knee during all visits (#1-13). Pain will be assessed with NRS (numeric rating scale) where 0 is no pain and 10 is worst possible pain.

SECONDARY OUTCOMES:
Changes in mobility | 12 weeks
  Mobility will be assessed via Timed Up & Go (TUG) assessment during visits #1, 12, 13. Participants are timed getting up from sitting in a standard armchair, walking approximately 3 meters, turning, walking back to the chair, and sitting down.
Changes in patient-relevant outcomes | 12 weeks
  Patient-relevant outcomes will be assessed via the Knee Injury and Osteoarthritis Outcome Score (KOOS) during visits #1, 12 and 13. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. KOOS does not use a numerical scale, it uses a qualitative scale with the following options: never, rarely, sometimes, often and always.
Changes in brief pain inventory | 12 weeks
  The brief pain inventory (BPI) will be used to assess changes in pain during visits #1, 12, and 13. This scale ranges from 0 to 10. The numerical value 0 can represent "no pain" or "does not interfere". The numerical value 10 can represent "pain as bad as you can imagine" or completely interferes".
Changes in the use of pain medication | 12 weeks
  Medication usage will be recorded during visits #1, 12, 13 and any increase/decrease in pain medications will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Thiru Annaswamy, MD, Principal Investigator — Veteran Affairs North Texas Healthcare System
Locations (1):
- Veteran Affairs North Texas Healthcare System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No